CLINICAL TRIAL: NCT01300689
Title: Human Papillomavirus Infection and Knowledge and Attitudes About HPV Vaccines Among Men Who Have Sex With Men (MSM)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Lei Gao, Institute of Pathogen Biology, Chinese Academy of Medical Sciences & Peking Union Medical College
Organization: ChineseAMS (Unknown)
Other Study IDs: HPV and MSM in China
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: HPV Infection; HIV Infection; Syphilis
Keywords: HPV; MSM; Vaccine; China
MeSH Terms: conditions — Papillomavirus Infections; HIV Infections; Syphilis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a observational study aims to assess anal and genital human papillomavirus (HPV) infection status among men who have sex with men (MSM) in China, and their knowledge and attitude about HPV vaccine.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old;
* Ever had homosexual behaviors in the past 12 months;
* Willing to take tests for HIV/HPV infection;
* Physically able and willing to provide written informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 3,000 eligible men who have sex with men (MSM) with 300 from each city will be enrolled from ten cities (BeiJing, ShangHai, TianJin, ChongQing, GuangZhou, ZhengZhou, Harbin, ShenYang, ChengDu, and KunMing) by the local CDCs and non-government MSM organizations
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2011-07

CONTACTS AND LOCATIONS:
Overall Officials: Lei Gao, Ph.D., Principal Investigator — Institute of Pathogen Biology (IPB), CAMS&PUMC
Locations (1):
- Institute of Pathogen Biology (IPB), Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Gao L, Zhou F, Li X, Yang Y, Ruan Y, Jin Q. Anal HPV infection in HIV-positive men who have sex with men from China. PLoS One. 2010 Dec 6;5(12):e15256. doi: 10.1371/journal.pone.0015256. PMID 21151900